CLINICAL TRIAL: NCT00353340
Title: Prevention of Contrast Nephropathy by Sodium Bicarbonate Versus Sodium Chloride and N-acetylcysteine in Patients Undergoing Cardiac Catheterization
Brief Title: Prevention of Contrast Nephropathy by Sodium Bicarbonate Versus Sodium Chloride and N-acetylcysteine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 70202
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Acute Renal Failure Contrast Nephropathy
Keywords: sodium bicarbonate,; n-acetylcisteine,; contrast nephropathy,; cardiac catheterisation
MeSH Terms: interventions — Acetylcysteine; Sodium Bicarbonate; Sodium Chloride

INTERVENTIONS:
Drug: n acetylcysteine
Drug: sodium bicarbonate
Drug: sodium chloride

SUMMARY:
The objective of this study is to assess the efficacy of sodium bicarbonate compared with sodium chloride and oral N-acetylcysteine (NAC ) pretreatment for prevention of contrast nephropathy in patients with advanced renal disease undergoing cardiac catheterisation.

DETAILED DESCRIPTION:
PROTOCOL

Prevention of Contrast Nephropathy by Sodium Bicarbonate Versus Sodium Chloride and N-Acetylcysteine

Nephrology and Cardiology Services, Shaare Zedek Medical Center, Jerusalem

1. Background and rationale

   The development of acute renal failure following cardiac catheterization has been recognized since the 1970's. The syndrome of acute renal failure following cardiac catheterization is presently felt to be due either to atheroembolic disease or what is now referred to as contrast induced nephropathy. Since the clinical course of each is different, it is now usually not difficult to diagnose acute contrast induced nephropathy.

   All protocols to prevent contrast nephropathy include the infusion of sodium chloride with or without oral N-acetylcysteine (NAC) pretreatment, although several recent meta-analyses raise some doubt about the efficacy of.

   Review of Shaare Zedek Medical Center experience from 2000 thru 2003 demonstrated a significant decrease in the incidence of acute contrast induced nephropathy after cardiac catheterization following the introduction of routine NAC usage. This effect was detected in a patients with mild renal insufficiency only (creatinine less than 1.5mg/dl). Patients with higher plasma creatinines did not appear to benefit from NAC prophylaxis.

   A recent study demonstrated that preventive hydration with sodium bicarbonate was more effective than sodium chloride in patients undergoing radiographic procedures. However, in that study, there was no subdivision of the patients by severity of their kidney disease and it is not clear if sodium bicarbonate was as effective in patients with more severe kidney disease as in those with milder renal impairment. In addition the rate, duration and kind of fluids that were used for preventive hydration differed from that currently recommended.

   Because free radicals are postulated to mediate contrast induced nephropathy and their formation is promoted by an acidic environment, alkalinizing renal tubular fluid with bicarbonate may reduce renal injury by reducing free radial formation. NAC is also known to be a free radical scavenger but since this compound was relatively ineffective in preventing contrast nephropathy in our patients with moderate to severe renal impairment (plasma creatinine > 1.5 mg%), we postulate that sodium bicarbonate may be more effective in the prevention of contrast nephropathy in these high risk patients.

   The proposed study is designed to test the efficacy of preventive hydration with sodium bicarbonate versus sodium chloride and oral NAC pretreatment in patients with stable advanced renal insufficiency (CKD stage 3 and 4-GFR 15-60ml/min/1.73m2 calculated by MDRD formula) undergoing cardiac catheterization.
2. Study objectives

   The objective of this study is to assess the efficacy of sodium bicarbonate compared with sodium chloride and NACpretreatment for prevention of contrast nephropathy in patients with advanced renal disease.
3. Outcome measure

   The incidence of contrast induced nephropathy, defined as 25% or more increase in serum creatinine within 2 days of contrast administration, will be assessed.
4. Study design

   This is a prospective, randomized, single center trial. Patients due to undergo cardiac catheterization either electively or following acute coronary syndromes will be eligible for inclusion. Elective patients will be admitted the day before the procedure. After baseline assessment and laboratory tests, they will be randomly assigned to one of two groups. One group will receive 12 hours infusion of 154 meq/l (0.9%) sodium chloride at a rate of 1ml/kg per hour before cardiac catheterization and NAC 600mg x 2/d PO the day before and the day of the procedure.

   The second group will receive 154meq/l sodium bicarbonate in 5% dextrose in water mixed by the nursing staff by adding 154 ml of 1000 meq/l sodium bicarbonate to 846 ml of 5% dextrose in water, slightly diluting the dextrose concentration to 4.23%.The initial IV bolus will be 3 ml/kg for one hour before cardiac catheterization. Following this bolus, patients will receive the same fluid at a rate of 1 ml/kg per hour during the contrast exposure and for 6 hours after the procedure.

   A basic panel of blood chemistries (Na, K, Cl, Ca, P, BUN, creatinine, total protein, albumin, complete blood count, pH, HCO3, pCO2 and O2 sat) will be obtained before the procedure and post-procedure day 1 and 2 and until any increase of serum creatinine is resolved. GFR will be calculated by MDRD formula in all patients before cardiac catheterization.
5. Patient selection

   Patients will be identified as study candidates based on preliminary laboratory tests results. They will referred from the clinics of Shaare Zedek, Kupot Cholim and the inpatient services of Shaare Zedek Medical Center. Eligible patients include individuals aged 18 year or older with GFR 15-60ml/min calculated by MDRD formula, who were scheduled to undergo cardiac catheterization. During the randomized study, consecutive eligible patients scheduled for exposure to the nonionic radiographic contrast agent iopamidol (796 mOsm/kg H2O, 755 mg of iopamidol per milliliter, and 370 mg iodine per milliliter) will be considered for enrollment.
6. Exclusion criteria

   i. Serum creatinine levels more than 8mg/dl or GFR less than 15ml/min

   ii. Change in serum creatinine levels of ³0.5mg/dl during the previous 24 hours.

   iii. Preexisting dialysis

   iv. Multiple myeloma.

   v. Pulmonary edema.

   vi. Uncontrolled hypertension (treated systolic blood pressure more than 160 mmHg, or diastolic blood pressure more than 100mmHg.)

   vii. Emergency catheterization.

   viii. Recent exposure to radiographic contrast (within two days of the study).

   ix. Allergy to radiocontrast.

   x. Pregnancy.

   xi. Administration of dopamine, mannitol or NAC before the study.
7. Blinding

   The study will be completely blinded. The serum creatinine level will be determined in a fully blinded fashion by laboratory personnel. The investigators from the Nephrology service will analyze the laboratory data without knowledge of patient study groups. The patients will not know to which group they will be randomized. The investigators from the Cardiology service will know the patient study groups, but will not analyze the patients laboratory tests results.
8. Study Methods

   Qualified patients who agree to enter the study will be assigned to 1 of 2 treatment groups based on a computer-generated randomization schedule. Patients allocated to the sodium chloride-NAC group will receive 154mEq/L of sodium chloride at a rate of 1ml/kg per hour for 12 hours before cardiac catheterization and NAC 600mgx2/d PO the day before and the day of the procedure. Patients allocated to the sodium bicarbonate group will receive 154 mEq/L of sodium bicarbonate in dextrose and H2O, mixed by the Nursing Service by adding 154 mL of 1000 mEq/L sodium bicarbonate to 846 mL of 5% dextrose in H2O, slightly diluting the dextrose concentration to 4.23%.

   After appropriate nursing evaluation and initial measurement of blood pressure and weight, the pre-contrast fluid will be administered. Patients allocated to the sodium chloride-NACgroup will receive 154 mEq/L of sodium chloride at a rate of 1ml/kg per hour for 12 hours before cardiac catheterization and NAC 600mgx2/d PO the day before and the day of the procedure The initial intravenous bolus in the NaHCO3 group will be 3 mL/kg per hour for 1 hour immediately before radiocontrast injection. Following this, patients will receive the same fluid at a rate of 1 mL/kg per hour during the contrast exposure and for 6 hours after the procedure. For patients weighing more than 110 kg, the initial fluid bolus and drip will be limited to those doses administered to a patient weighing 110 kg. Diuretics will be routinely withheld on the day of contrast injection. A basic panel of blood chemistries (Na, K, Cl, Ca, P, BUN, creatinine, total protein, albumin, complete blood count, serum pH, HCO3, pCO2 and O2 sat)) will be obtained before the procedure and post-procedure days 1 and 2 and until any increase of serum creatinine is resolved. GFR will be calculated by MDRD formula before the procedure.
9. Study End Points and Statistical Analysis

   The primary outcome measure is development of contrast-induced nephropathy, defined by an increase in serum creatinine of 25% or more within 2 days after cardiac catheterization. This definition is identical to that used in a recent large meta-analysis in contrast-induced nephropathy. Post-contrast creatinine will be assessed the mornings of days 1 and 2. The highest serum creatinine on post-contrast days 1 or 2 will be used to calculate the change in serum creatinine (the primary end point).

   Before beginning the study, we estimated the sample size needed for the primary end point of contrast-induced nephropathy. Based on our own and other previous data, we assumed the development of contrast-induced renal failure in 15% of the sodium chloride-NAC group and 5 % of the sodium bicarbonate group. Analysis indicated that a sample size of 281 patients would be required to detect a statistically significant difference with a power of 80% (two tailed p = 0.05).

   Tests for significance will be conducted using the t test for continuous variables and c2 or Fisher exact test for categorical variables. All analyses will be conducted using SAS software version 8.2 (SAS Institute Inc, Cary, NC). Data will be expressed as mean (SD). All tests will be 2-tailed, with differences reported as significant if p <0.05.
10. Feasibility of the study

    The average number of cardiac catheterizations performed in Shaare Zedek Medical Center is 25-30 procedures per week. A recent review of 30 consecutive cardiac catheterization patients showed that 8 would be eligible for enrollment in this protocol. Thus, it should take about 10-12 months to enroll the required number of patients.
11. Safety

    The infusion of sodium bicarbonate and sodium chloride is safe. In the published sodium bicarbonate study bolus administration of hydration fluids caused a moderate increase in both systolic and diastolic blood pressure (mean 11mm Hg in the sodium chloride group and 14 mmHg in the sodium bicarbonate group.) No patients developed clinical heart failure or respiratory distress. Since the patients enrolled in our study should have controlled hypertension (patients with blood pressure more than 160/100 will be excluded) this mild elevation in blood pressure should not be problematic.
12. Study significance

Contrast induced nephropathy is a common complication of cardiac catheterizations. Prophylactic hydration with sodium chloride and NAC which is currently in use is less effective in patients with advanced renal disease and the observed incidence of acute contrast induced nephropathy is approximately 15%. In addition the use of this regimen requires preventive hospitalization and may be especially problematic in patients with chronic kidney disease when they require urgent cardiac catheterization. If preventive hydration with sodium bicarbonate is as effective or better than the currently used saline-NAC regimen, the pretreatment time for cardiac catheterization could be significantly shortened, hence permitting its usage before emergent procedure. Since emergent procedures preclude the use of current relatively long pretreatment regimens, bicarbonate could reduce the incidence of acute contrast induced nephropathy in this highly vulnerable group.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients include individuals aged 18 year or older with GFR 15-60ml/min calculated by MDRD formula, who were scheduled to undergo cardiac catheterization. During the randomized study, consecutive eligible patients scheduled for exposure to the nonionic radiographic contrast agent iopamidol (796 mOsm/kg H2O, 755 mg of iopamidol per milliliter, and 370 mg iodine per milliliter) will be considered for enrollment.

Exclusion Criteria:

i. Serum creatinine levels more than 8mg/dl or GFR less than 15ml/min

ii. Change in serum creatinine levels of ³0.5mg/dl during the previous 24 hours.

iii. Preexisting dialysis

iv. Multiple myeloma.

v. Pulmonary edema.

vi. Uncontrolled hypertension (treated systolic blood pressure more than 160 mmHg, or diastolic blood pressure more than 100mmHg.)

vii. Emergency catheterization.

viii. Recent exposure to radiographic contrast (within two days of the study).

ix. Allergy to radiocontrast.

x. Pregnancy.

xi. Administration of dopamine, mannitol or NAC before the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The incidence of contrast induced nephropathy, defined as 25% or more increase in serum creatinine within 2 days of contrast administration, will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: linda shavit, md, Principal Investigator
Locations (1):
- Shaare Zmc, Jerusalem, Israel